CLINICAL TRIAL: NCT00070863
Title: Behavior Therapy for Partner Violent Men
Brief Title: Treatment for Men Who Are Abusive to Their Partners
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore County (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Timothy A Sparklin, Research Compliance Officer, University of Maryland, Baltimore County
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21MH064562 (NIH); R21MH064562 (NIH); DSIR AT-AS
Record Dates: First submitted 2003-10-08; First posted 2003-10-09 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Domestic Violence

INTERVENTIONS:
Behavioral: Individual Cognitive Behavioral Therapy

SUMMARY:
This study will develop an individual behavior therapy for men who are violent toward their partners and will compare the therapy to standard group treatment.

DETAILED DESCRIPTION:
To date, treatment interventions for domestic abuse perpetrators have been conducted almost exclusively in groups. However, the efficacy of such treatments relative to no treatment has not been thoroughly evaluated. Evidence suggests that individual treatments may be more effective than group treatments. This study will combine motivational enhancement therapy with cognitive and behavior change techniques to treat men who abuse their partners.

This study will be conducted in two phases. In Phase 1, an individual cognitive behavior therapy (ICBT) manual will be constructed. During Phase 2, participants will be randomly assigned to receive either 16 sessions of ICBT or 16 sessions of standard group therapy. Data on abusive behavior outcomes and secondary treatment targets will be collected from participants and their partners every 3 months for 1 year after the study.

ELIGIBILITY:
Inclusion Criteria:

* Involved in male-to-female physical aggression in the past 12 months or has a history of severe male-to-female aggression in a relationship
* Current involvement in a primary intimate relationship (cohabiting, dating, or married) for at least 6 months, with partner contact at least once per week
* Willingness to provide written consent for partner contact
* Partner provides verbal assent for the use of information during an initial phone interview and agrees to be re-contacted for scheduled follow-up interviews

Exclusion Criteria:

* Psychotic symptoms or severe mood disorder
* Mental retardation, autism, dementia, delirium, catatonia, or other severe cognitive disorders
* Severe head trauma in the past two years
* Seizure disorder
* Current diagnosis of alcohol dependence or drug dependence. Participants must be in remission for at least 6 months if a past diagnosis is present.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-06; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Individual Versus Group Cognitive-Behavioral Therapy for Partner-Violent Men study of physical assault, emotional abuse, and injury as reported by the male participant and his relationship partner | Three month intervals for one year after the initiation of treatment
  Physical assault, emotional abuse, and injury as reported by the male participant and his relationship partner

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M. Murphy, PhD, Principal Investigator — University of Maryland, Baltimore County
Locations (1):
- Domestic Violence Center of Howard County, Columbia, Maryland, United States